CLINICAL TRIAL: NCT07391345
Title: A Prospective, Randomized, Three-Arm, Open-Label Clinical Trial Comparing Transoral CO₂ Laser Microsurgery, Volumetric Modulated Arc Therapy (VMAT), and MRI-Guided Stereotactic Ablative Radiotherapy (MRI-SABR) in the Treatment of Early-Stage Glottic Laryngeal Cancer
Brief Title: Precision Medicine: MRI-Guided Stereotactic Ablative Radiotherapy (MRI-SABR) for Early-Stage Glottic Laryngeal Cancer
Acronym: SMART - 1_1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Viktoras Rudzianskas (Other)
Responsible Party: Sponsor-Investigator, Viktoras Rudzianskas, Principal investigator, Associate professor, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE-2-45
Record Dates: First submitted 2026-01-15; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Laryngeal Neoplasm; Glottic Carcinoma
Keywords: Early-stage glottic laryngeal cancer; transoral laser microsurgery; VMAT; MRI-SABR; stereotactic radiotherapy; radiomics; dosiomics
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Transoral CO₂ Laser Microsurgery (TLM) (Active Comparator): Participants undergo transoral CO₂ laser microsurgery for the treatment of early-stage glottic laryngeal cancer.
  Interventions: Procedure: Transoral CO₂ laser cordectomy (Type I-VI depending on tumor localization)
- Arm B: Volumetric Modulated Arc Therapy (VMAT) (Active Comparator): Participants receive definitive external beam radiotherapy using volumetric modulated arc therapy.
  Interventions: Radiation: VMAT radiotherapy
- Arm C: MRI-Guided Stereotactic Ablative Radiotherapy (MRI-SABR) (Active Comparator): Participants receive definitive MRI-guided stereotactic ablative radiotherapy.
  Interventions: Radiation: MRI-SABR

INTERVENTIONS:
Procedure: Transoral CO₂ laser cordectomy (Type I-VI depending on tumor localization) — Surgical removal of the tumor with at least 2 mm margins; intraoperative frozen section biopsies; short hospitalization (1-3 days).
  Arms: Arm A: Transoral CO₂ Laser Microsurgery (TLM)
Radiation: VMAT radiotherapy — Accelerated fractionation schedule: T1N0 - 63 Gy/28 fractions; T2N0 - 65.25 Gy/29 fractions; delivered using Eclipse planning system.
  Arms: Arm B: Volumetric Modulated Arc Therapy (VMAT)
Radiation: MRI-SABR — 42.5 Gy total dose in 5 fractions, 2 fractions per week, planned with CT and MRI simulation and delivered with MRI-LINAC system.
  Arms: Arm C: MRI-Guided Stereotactic Ablative Radiotherapy (MRI-SABR)

SUMMARY:
This randomized phase III trial will compare the outcomes of three treatment modalities for early-stage glottic laryngeal cancer (T1-T2N0): transoral CO₂ laser microsurgery (TLM), volumetric modulated arc therapy (VMAT), and MRI-guided stereotactic ablative radiotherapy (MRI-SABR). The primary endpoint is local control (LC). Secondary endpoints include laryngectomy-free survival (LFS), progression-free survival (PFS). overall survival (OS), functional voice, swallowing and breathing outcomes, treatment-related complications, and the evaluation of radiomic and dosiomic biomarkers. Patients will be randomized in a 1:1:1 ratio. Total planned enrollment is 105.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Histologically confirmed squamous cell carcinoma of the glottic larynx, including verrucous carcinoma.
* Stage T1-T2N0 (8th TNM edition).
* ECOG performance status 0-2.
* Able to understand Lithuanian and complete questionnaires.
* Signed informed consent.

Exclusion Criteria:

* AJCC stage III-IV laryngeal cancer.
* Prior radiotherapy for head and neck cancer.
* Pregnancy or breastfeeding.
* Contraindications for radiotherapy or inability to follow-up.
* Presence of another active malignancy.
* Uncontrolled intercurrent illness (e.g., active infection, symptomatic CHF, unstable angina, clinically significant arrhythmia) or any condition that would preclude radiotherapy or adequate follow-up per investigator judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Local Tumor Control Rate Assessed by Endoscopy and Imaging | At 2 years after completion of treatment; At 5 years after completion of treatment
  Proportion of participants without local tumor recurrence, assessed by laryngoscopic examination and radiological imaging.

SECONDARY OUTCOMES:
Laryngectomy-Free Survival (LFS) | Up to 2 years after randomization; Up to 5 years after randomization
  Time from randomization to total laryngectomy or death from any cause, whichever occurs first.
Progression-Free Survival (PFS) | Up to 2 years after randomization; Up to 5 years after randomization
  Time from randomization to disease progression (local, regional, or distant) or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 years after randomization; Up to 5 years after randomization
  Time from randomization to death from any cause.
Objective Voice Parameters Assessed by Acoustic Analysis (lingWAVES) | Baseline, and at 1, 3, 6, 12, 18, and 24 months after completion of treatment
  Objective voice parameters derived from acoustic signal analysis using the lingWAVES system.
Patient-Reported Voice Outcome Assessed by Voice Screen Application | Baseline, and at 1, 3, 6, 12, 18, and 24 months after completion of treatment
  Patient-reported voice outcome assessed using the Voice Screen mobile application.
Swallowing Function Score Assessed by Anderson Dysphagia Inventory | Baseline, and at 1, 3, 6, 12, 18, and 24 months after completion of treatment
  Swallowing function assessed using the Anderson Dysphagia Inventory questionnaire (total score).
Health-Related Quality of Life Scores Assessed by EORTC QLQ-C30 and QLQ-H&N35 | Baseline, and at 1, 3, 6, 12, 18, and 24 months after completion of treatment
  Health-related quality of life assessed using the EORTC QLQ-C30 and QLQ-H&N35 questionnaires (global health status and domain scores).
Quantitative Radiomic and Dosiomic Feature Values and Their Statistical Associations With Clinical Outcomes | From baseline imaging through 5 years after completion of treatment
  Quantitative radiomic feature values extracted from baseline and follow-up imaging (CT, MRI, PET/CT) and quantitative dosiomic feature values derived from radiotherapy treatment plans. Associations with clinical outcomes (local tumor control, progression-free survival, overall survival) will be summarized using correlation coefficients and hazard ratios.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No